CLINICAL TRIAL: NCT07225998
Title: The NAGIC Study: Multi-center, Randomized, Double-blind, Placebo-controlled Cross-over Study of Oral N-acetylglucosamine in Ileal/Ileocolonic Crohn's Disease
Brief Title: Oral N-acetylglucosamine in Crohn's Disease
Acronym: NAGIC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Leona M. & Harry B. Helmsley Charitable Trust (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00533883; R01DK141870 (NIH); 2604-09127 (Other Grant/Funding Number: Leona M. & Harry B. Helmsley Charitable Trust)
Record Dates: First submitted 2025-10-29; First posted 2025-11-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Crohns Disease
Keywords: Crohns disease; manganese; GlcNAc; N-acetylglucosamine; ZIP8 protein; SLC39A8 gene; genetics; glycosylation disorder
MeSH Terms: conditions — Crohn Disease | interventions — Acetylglucosamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with Crohn's disease and carry ZIP8 391-Thr (heterozygous or homozygous carriers) (Experimental): N-acetylglucosamine
  Interventions: Drug: N-Acetylglucosamine (GlcNAc)
- Participants with Crohn's disease who do not carry ZIP8 391-Thr (Experimental): N-acetylglucosamine
  Interventions: Drug: N-Acetylglucosamine (GlcNAc)

INTERVENTIONS:
Drug: N-Acetylglucosamine (GlcNAc) — This is a placebo-controlled, cross-over design. The sequence in which the participant receives the GlcNAc or placebo is randomized. Participants will take GlcNAc 2 grams three times daily or placebo (glucose 2 grams three times daily) for 6 weeks. There will then be a 3 week washout period and then cross-over to GlcNAc or placebo for 6 weeks. Participants will be followed for 3 weeks off all drug/placebo to complete the study at week 18.

SUMMARY:
Protein glycosylation is a critical post-translational modification that regulates protein trafficking and protein-protein interactions impacting a host of physiological processes. There is a growing appreciation of glycosylation defects in chronic human diseases, including Crohns disease. Crohns disease (CD), and the related condition of ulcerative colitis, are chronic inflammatory bowel diseases (IBD) that impact 3.1 million Americans. While the development of medications has revolutionized care of CD patients, clinical remission is only achieved in ~40% of patients a therapeutic ceiling that has not changed in 20 years. These data underscore the need for new CD treatment strategies. The investigators are focused on understanding the role of defective N-glycosylation in CD, as an innovative strategy to identify and develop new therapeutics. Depending on ancestral background, 7-25% of CD patients carry a pathogenic, missense mutation in the manganese (Mn) transporter ZIP8 (rs13107325; ZIP8 A391T). ZIP8 regulates systemic Mn homeostasis with ZIP8 391-Thr causing a relative Mn insufficiency. Mn is a required metal cofactor for enzymes regulating key cellular processes, like N-glycosylation. In the gut, protein N-glycosylation plays key roles in host-pathogen interactions, inflammation, and cell-cell interactions. The investigator's central hypothesis is that in patients carrying ZIP8 391-Thr - CD is exacerbated by aberrant N-glycosylation and that this defect can be targeted by specific, safe therapy. Supporting this hypothesis, Mn levels are reduced (~15%) in ZIP8 391-Thr allele carriers and this is associated with a decrease in complex N-glycan branching in plasma. Further, the investigators uncovered a microbiota signature in the ileal mucosa that implicated altered bile acid homeostasis in ZIP8 391-Thr carriers. To better understand CD in ZIP8 391 carriers, the investigators generated a knock-in mouse model of ZIP8 391-Thr (Zip8393T/393T). Like patient data, the investigators observe reduced branching of N-glycans and disrupted bile acid homeostasis in the Zip8393T/393T mice. Promising human trials have shown that defects in N-glycan branching can be safely restored by raising levels of the rate-limiting metabolite UDP-N-acetylglucosamine (GlcNAc) via supplementation with free GlcNAc. The investigator's preliminary data in Zip8393T/393T mice have demonstrated that GlcNAc supplementation restores N-glycan branching deficits, rescues the defect in bile acid homeostasis, and ameliorates colitis susceptibility. Thus, the objective of the proposed research is to test a safe and effective therapy for patients carrying ZIP8 391-Thr and others who may have underlying changes in N-glycosylation.

The investigators will perform a multi-center, randomized, double-blind, placebo-controlled cross-over study to test the safety and tolerability of oral GlcNAc as a proof-of-concept study. The investigators will use two cohorts stratified by ZIP8 391-Thr genotype status (carriers and non-carriers, n= 20 participants in each cohort, total= 40 participants).

DETAILED DESCRIPTION:
While many new medications improved care for patients with Crohn's disease, clinical remission is only achieved in ~40% of patients - a therapeutic ceiling that has not changed in 20 years. These data underscore the need for new treatment strategies and (the investigators hypothesize) greater focus on personalized medicine using factors like genetics.

This study is a clinical trial of oral N-acetylglucosamine (GlcNAc) in patients with Crohn's disease. The investigators are aiming for approximately half of the participants to carry a genetic variant in a gene called ZIP8. ZIP8 regulates levels of manganese and the variant lowers levels of manganese; manganese levels may also be reduced for reasons other than just ZIP8 genetics - including variation in dietary intake, water sources, and inflammation - therefore, the investigators are also enrolling participants who do not have the ZIP8 variant. Manganese is a nutrient absorbed from food that is required for glycosylation, but direct supplementation of excess manganese may carry risk of neurologic side effects. An alternative approach is to supplement with GlcNAc, the critical building block of glycosylation that regulates intestinal health and inflammation. GlcNAc is preferred given its positive safety profile and prior small studies in patients with inflammatory bowel disease that showed promising results.

Key study information:

* The investigators will check if the participant carries the ZIP8 variant at study enrollment. The participants can choose to be informed of ZIP8 genetics.
* This is a randomized, double-blind, placebo-controlled, cross-over study. This study design provides the most power to determine if there is a beneficial effect of GlcNAc.
* This means the participant will receive the study drug (GlcNAc), but will also have a period of placebo. The sequence in which the participant receives the GlcNAc or placebo is randomized. The study is blinded, meaning that the participant and the investigator will not know if the participant is receiving active drug or placebo unless there are safety concerns.
* GlcNAc or placebo is provided to the participant as a powder that the participant will mix in a small amount of water 3 times per day.
* GlcNAc is a naturally-occurring substance found in nature and tastes sweet when mixed with water.
* The study runs for 18 weeks. There are brief, weekly check-ins and 7-8 in-person visits.
* Participants will be asked to provide blood, stool, and saliva samples for a total of 7-8 times.
* If it is possible at the participant's site, intestinal ultrasounds will be performed over the course of the study.

  * Participants will be paid to participate in the study. There are no direct costs to the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and 80 years of age
2. Diagnosis of CD involving ileum (L1) or ileocolonic disease (L3) of any disease behavior
3. On stable dosing of any CD therapy for >/= 8 weeks (inclusive of biologics, small molecules, immunomodulators)
4. CDAI <450
5. Willing to undergo genetic testing for ZIP8 genotype
6. No steroids within the past 4 weeks
7. No antibiotics within the past 2 weeks
8. Willing to provide informed consent
9. Willing to participate in all at-home and clinic-based follow-up
10. Willing to provide most recent endoscopy and imaging results; when possible, access to prior pathology specimens
11. Willing to use all forms of "highly effective" contraception throughout the study period and for 30 days after the last dose of study drug (all subjects of child-bearing potential)

Exclusion criteria

1. Have taken GlcNAc or glucosamine in the previous 3 months
2. Allergy to shellfish
3. Severely-active CD defined as CDAI >450 AND/OR
4. Simple Endoscopic Score for Crohn's Disease (SES-CD) score >/= 16 (or >/= 8 for isolated ileitis) on colonoscopy within 8 weeks of screening, if available
5. Steroids within the past 4 weeks
6. Antibiotics within the past 2 weeks
7. Stricture with high-grade obstruction, significant fistulizing disease, presence of intra-abdominal or perianal abscess, perforation, or fulminant colitis requiring imminent surgical management
8. Surgery within 12 weeks
9. Recent initiation or escalation of immunosuppressive therapy (<8 weeks)
10. Any clinically significant abnormalities on routine clinical labs, including unexplained white blood cells (WBC) >16,000, hemoglobin <7, AST/ALT >2x ULN, alkaline phosphatase >2x ULN, eGFR <60, ferritin <30 ng/ml2
11. History of type 1 diabetes, inadequately controlled type 2 diabetes (HbA1c>6.5%), type 2 diabetes on insulin
12. History of peripheral vascular disease, coronary artery disease, stroke, transient ischemic attack
13. History of cancer
14. History of organ transplant
15. History of bleeding disorder
16. History of chronic respiratory disorder, including asthma
17. History of chronic renal failure
18. History of chronic liver disease, including primary sclerosing cholangitis
19. History of seizure disorder
20. Pregnant, less than 6 months postpartum, breastfeeding, or attempting to conceive

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: Number of Crohn's disease exacerbations | Weeks 0-6, Weeks 6-9, Weeks 9-15, Weeks 15-18
  Safety and tolerability will be defined as freedom from Crohn's disease (CD) disease exacerbation. Number of CD exacerbations will be one composite outcome with exacerbation of CD activity defined as the occurrence of ANY of the following during each treatment phase:
  i. Crohn's disease activity index (CDAI) score (patient reported measure) change of >100 points, ii. initiation or change of CD therapy due to symptom worsening, iii. need for steroids related to CD disease activity, iv. CD-associated hospitalization, v. CD-associated surgery, vi. severe adverse events (CTCAE grade 3-5, attributed to CD disease activity, e.g. life-threatening perforation or sepsis)

SECONDARY OUTCOMES:
Clinical response as assessed by CDAI score | Week 6, week 15 for each treatment phase (GlcNAc and placebo)
  Patient reported disease activity index: CDAI score range from 0 to 600; scores <150 define remission, 150 to 219 mild activity, 220 to 450 moderate activity, and greater than 450 severe activity.
  Clinical response will be defined as a ≥70 point reduction in CDAI score from baseline by the end of the six-week treatment period stratified by disease activity at week 0.
Clinical response as assessed by mean change in CDAI score | Week 6, week 15 for each treatment phase (GlcNAc and placebo).
  Patient reported disease activity index: CDAI score range from 0 to 600; scores <150 define remission, 150 to 219 mild activity, 220 to 450 moderate activity, and greater than 450 severe activity. Within-participant change from baseline in CDAI score stratified by disease activity at week 0.
Clinical remission as assessed by CDAI score | Week 6, week 15 for each treatment phase (GlcNAc and placebo).
  Patient reported disease activity index: CDAI score range from 0 to 600; scores <150 define remission, 150 to 219 mild activity, 220 to 450 moderate activity, and greater than 450 severe activity. Clinical remission will be defined as a CDAI score of <150 at the end of the six-week treatment period stratified by disease activity at week 0.
Change in serum N-glycome | Week 0, 6, 9, 15, 18
  Measure of glycosylation Serum N-glycome (%): Change in Serum N-glycome from baseline to follow-up
Change in saliva N-glycome | Week 0, 6, 9, 15, 18
  Measure of glycosylation: Change in saliva N-glycome (%) from baseline to follow-up.
Mean change in serum UDP-GlcNAc | Week 0, 6, 9, 15, 18
  Measure of glycosylation: Serum UDP-GlcNAc (uM). Mean change in serum UDP-GlcNAc from baseline to follow-up.
Change in T cell N-glycan branching | Week 0, 6, 9, 15, 18
  Measure of glycosylation: Change in T cell N-glycan branching (%) from baseline to follow-up
Change in T cell activity/responsiveness | Week 0, 6, 9, 15, 18
  Measure of glycosylation: Change in T cell activity/responsiveness (%) from baseline to follow-up
Change in fecal mucins | Week 0, 6, 9, 15, 18
  Measure of glycosylation: Change in fecal mucins (%) from baseline to follow-up
Mean change in fecal calprotectin | Week 0, 6, 9, 15, 18
  Measure of inflammation. Mean change in fecal calprotectin (%) from baseline to follow-up
Mean change in serum C-Reactive Protein (CRP) | Week 0, 6, 9, 15, 18
  Measure of inflammation: CRP (ng/ml) from baseline to follow-up
Change in panel-based blood inflammatory cytokines | Week 0, 6, 9, 15, 18
  Measure of inflammation: Change in panel-based blood inflammatory cytokines (pg/ml) measures from baseline to follow-up.
Change in marker of bile acid homeostasis (FGF19) | Week 0, 6, 9, 15, 18
  FGF19 is a circulating protein that is a marker of bile acid homeostasis.
Mean change in sCD14 | Week 0, 6, 9, 15, 18
  Measure of intestinal permeability sCD14 (pg/ml). Mean change in sCD14 from baseline to follow-up.
Mean Change in FACIT-Fatigue Patient-reported measure (Fatigue) | Week 0, 6, 9, 15, 18
  Patient-reported measure. Mean change in FACIT-Fatigue scores from baseline (Week 0) to final intervention (Week 13), with a clinical significant threshold set at >/= 4 points. Score ranges from 0 to 52 with higher scores indicating worse fatigue.
Mean Change in Simple Ultrasound Activity (SUS-CD) Score Disease activity measured by intestinal ultrasound | Week 0, 6, 9, 15, 18
  Disease activity: Mean change in simple ultrasound activity score (includes bowel wall thickness and color Doppler signals) for Crohn's disease at Week 13. Score range 0-5 with 0-1 indicating normal or very mild disease; 2-3 moderate disease; 4-5 severe active disease.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Melia, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) (data collected for each person, including demographics, Crohn's disease history, lab results, adverse events) will be shared after publication of results for research collaborations. IPD will be shared as a deidentified dataset with no protected health information (PHI) as per Institutional Review Board (IRB) regulations. Data sharing agreement will be required.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available approximately 18 months after trial completion (after publication of results) and available for at least 5 years.
Access Criteria: Individuals interested in access the IPD and supporting information will be able to access data collected for each person, including demographics, Crohn's disease history, lab results, adverse events, after data use agreement is signed by relevant parties.

REFERENCES:
- [Background] Salvatore S, Heuschkel R, Tomlin S, Davies SE, Edwards S, Walker-Smith JA, French I, Murch SH. A pilot study of N-acetyl glucosamine, a nutritional substrate for glycosaminoglycan synthesis, in paediatric chronic inflammatory bowel disease. Aliment Pharmacol Ther. 2000 Dec;14(12):1567-79. doi: 10.1046/j.1365-2036.2000.00883.x. PMID 11121904
- [Background] Tomar V, Kang SD, Lin R, Brant SR, Lazarev M, Tressler C, Glunde K, Zachara N, Melia J. Aberrant N-glycosylation may be a therapeutic target in carriers of a common and highly pleiotropic variant in the manganese transporter ZIP8. HGG Adv. 2026 Jan 15;7(1):100517. doi: 10.1016/j.xhgg.2025.100517. Epub 2025 Sep 16. PMID 40963256